CLINICAL TRIAL: NCT00977847
Title: Integrating Patient Generated Family Health History From Varied Electronic Health Record Entry Portals
Brief Title: Integrating Patient Generated Family Health History From Varied Electronic Health Record (EHR) Entry Portals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jennifer S. Haas, MD, MSPH, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009P0011908; 1RC1HG005331-01 (NIH)
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Family Characteristics; Health Status; Family Research
Keywords: Family History; Electronic Health Record

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Interactive Voice Response Practice (Experimental): The introductory letter to patients will allow them an opportunity to "opt-out" of the study using a toll-free number. If they do not opt-out within 2 weeks of receiving the letter, the IVR system will make up to 15 call attempts over a 2 week period to reach the patient. The system will make outbound calls during preset hours. The system continuously checks the call list for the next scheduled call. Once contact is made, the spoken script greets the patient by name, authenticates identify, and will ask the patient the programmed questions. The IVR server will send completed family history assessments to the patients EHR as an HL7 compliant summary note as well as transmitting the separate coded responses for each condition/ family member to coded family history fields in the EHR.
  Interventions: Other: Electronic Health Portals for collecting Family History data
- Wireless Tablet PC Practice (Experimental): Patients will receive an info letter in advance of their visit explaining the project with description of what information they will be asked to provide. Study staff will train the practice staff to hand out and collect the tablets for the patient. Staff will be trained to verify a patient's identity to ensure that the family history is sent to the correct EHR record. The initial screen of the tablet PC portal will include a paragraph of informed consent, and patients in this practice will be given the opportunity to decline participation. For patients who participate, the completed family history data will be transmitted to the patient's EHR as an HL7 compliant note and transmitting separate coded responses for each condition/ family member to coded family history fields.
  Interventions: Other: Electronic Health Portals for collecting Family History data
- Internet Portal Practice (Experimental): Patients in this practice will receive the informational letter either by email or mail one month before their scheduled visit. It will have directions to access the MFHP website and how to transfer data through the hospitals secure internet portal (Patient Gateway). About 1/3 of patients are signed up to use this service. Those who do not have a Patient Gateway account will be provided with directions on how to establish this service. Patients will be required to have a Gateway account to ensure that the MFHP data file is sent securely to the correct EHR record. Patients in this arm will receive an initial email or letter with a single follow-up reminder sent 2 weeks later. For patients who participate, the completed family history data will be transmitted to the patient's EHR.
  Interventions: Other: Electronic Health Portals for collecting Family History data
- Usual Care Physician Assesment Practice (Active Comparator): Usual standard family history assessments will be conducted by physicians during the patient visit. This arm will allow us to account for any temporal trends in family history assessment.
  Interventions: Other: Electronic Health Portals for collecting Family History data

INTERVENTIONS:
Other: Electronic Health Portals for collecting Family History data — Comparison of multiple portals for integrating patient generated family history data into the electronic health record.

SUMMARY:
In the 21st century, the importance of family health history will increase as it will be essential to put detailed personal genetic information into the context of an individual's health, namely the context of how the shared code has played out in an individual and his/her closest relatives. These scientific developments in the investigators' understanding of genetics will demand a more comprehensive family history dataset for all patients, and the time limitations on healthcare providers demand a technology-driven solution that integrates an individual's knowledge of their family history with the medical records maintained by their health care providers. A solution does not currently exist by which most Americans can organize their family health history and then place it into their electronic health record (EHR). The investigators propose to develop and compare three different ways of proactively collecting family history information from patients using computer technology independent of a health care visit, including telephone (interactive voice response technology), tablet computers in a physician's waiting room, and a secure internet portal at home. These tools will be based on the US Surgeon General's My Family Health Portrait, an electronic family history collection tool. Family history data will be transferred and integrated with a patient's EHR in a large primary care network. This project will seek to demonstrate that family history data can be accurately reported by diverse patients using these technologies, and that these data can be integrated to tailor an individual's health care based on their familial risk.

DETAILED DESCRIPTION:
Background: The long established wisdom of including family health history as a key part of an individual's medical record has been invigorated by the new emphasis on personalized medicine. While in the past, family health history was used to understand an individual's disease risk and to focus disease prevention efforts, in 21st century medicine, family health history's importance will increase as it will be essential to put detailed personal genetic information into a clinical context, namely the context of how the shared code has played out in a person's closest relatives. This new need for family health history will demand a more comprehensive family history dataset for all patients, and the time limitations faced by healthcare providers demand a technology-driven solution whereby the patient performs primary data entry and the provider then refines these data. Solutions do not currently exist by which most Americans can organize their family health history and then place it into their electronic health record (EHR). My Family Health Portrait (MFHP) is an open source, electronic family history collection tool developed by the Surgeon General that offers interoperability with EHRs, yet to our knowledge has not been widely integrated because of limitations in the capacity of many EHRs to accept these data, and barriers to the systematic collection of these data in clinical practice. Additionally, obstacles exist for those individuals who are not computer literate or do not have access to a home computer. In order to capture patient-generated family history data across diverse patient populations, EHR's may need to offer patients a variety of data entry options which allow for differences in preference, convenience, computer literacy, and computer availability. This proposal seeks to develop new resources for family history data entry into the EHR. These resources will be developed, tested and validated in a primary care setting within of a large complex healthcare system.

Research Plan: The proposed project will examine the reach, effectiveness, adoption and implementation of three innovative portals to transfer and integrate patient generated family history data with an EHR.

Specific Aim 1 (technical development) is to develop the three portals for entry of patient generated family history data integrated with an EHR. The pathways will include: : (1) computer tablets in waiting rooms to complete the MFHP, (2) a secure internet portal to transfer data collected by patients at home using MFHP, and (3) an interactive voice response (IVR) system to collect the necessary data elements by phone. Each of these modalities will interface with the EHR of a large health delivery system using current data standards. Each of these modalities will be designed to interface with the EHR of a large health delivery system using current data standards using current data standards.

Specific Aim 2 (content development and validation) is to evaluate facilitators and barriers to the adoption, and implementation of these three electronic portals by assessing differences in patient preferences, privacy concerns, convenience, and understanding. The validity of the family history data collected by each of these three portals will also be assessed by a genetic counselor.

Specific Aim 3 (pilot randomized controlled trial) is to conduct a 4-armed pilot randomized controlled trial (RCT) to measure the reach and effectiveness of integrating this family history data with a patient's EHR. The trial will examine and compare changes in family history documentation, patient-doctor discussion of family history, and patient and provider satisfaction with each data entry portal described in Aim 1, as well as a control arm. The trial will be conducted as a pilot cluster RCT in selected practices within the Brigham and Women's Primary Care Practice-Based Research Network.

Potential Impact: The impact of obtaining accurate family history data and integrating this with an individual's health record are substantial, and will be of growing importance as our understanding of the genome advances. This project will ultimately contribute to a better understanding of how available technologies can be integrated with EHR's to obtain accurate family history in ways that allow for widespread acquisition and integration of accurate family history data in a variety of settings and diverse patient populations. The technology and lessons learned from this project will be exportable to healthcare settings throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

Male and Female Patients who:

* receive primary care at one of the study selected Primary Care Practices,
* are between 18-75 years old,
* are English or Spanish speakers, and
* have appointments scheduled in the upcoming 1 - 3 months for an annual or comprehensive visit.

Exclusion Criteria:

* We will not include individuals over the age of 75 because the role of family risk assessment and prevention is less established.
* Also will not include non-English or non-Spanish speakers.
* Patients will also be excluded if they are hearing impaired.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Project will seek to demonstrate that family history data can be accurately reported by 5000 diverse patients using three portals, and that these data can be used to tailor an individual's health care based on their familial risk. | 2.5 years

SECONDARY OUTCOMES:
Develop three portals for collection of patient generated family history data integrated with an EHR: computer tablets in waiting rooms; a secure internet portal for use at home; and an interactive voice response system to get data by phone. | 1.5 years
Evaluate facilitators and barriers to adoption and implementation of these portals by assessing differences in patient preferences, privacy, convenience, and understanding. Validate data collected by each portal by a genetic counselor. | 1.5 years
To conduct a 4-armed pilot RCT to measure the reach and effectiveness of integrating family history data with a patient's EHR. | 2 years
For patients in the RCT who report a family history that is associated with an increased risk of coronary artery disease, we will examine how often their physician initiates screening and/ or primary prevention based on the family history information. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Haas, MD, MSPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Yoon PW, Scheuner MT, Peterson-Oehlke KL, Gwinn M, Faucett A, Khoury MJ. Can family history be used as a tool for public health and preventive medicine? Genet Med. 2002 Jul-Aug;4(4):304-10. doi: 10.1097/00125817-200207000-00009. No abstract available. PMID 12172397
- [Background] Sabatino SA, McCarthy EP, Phillips RS, Burns RB. Breast cancer risk assessment and management in primary care: provider attitudes, practices, and barriers. Cancer Detect Prev. 2007;31(5):375-83. doi: 10.1016/j.cdp.2007.08.003. Epub 2007 Nov 26. PMID 18037249
- [Background] Acheson LS, Wiesner GL, Zyzanski SJ, Goodwin MA, Stange KC. Family history-taking in community family practice: implications for genetic screening. Genet Med. 2000 May-Jun;2(3):180-5. doi: 10.1097/00125817-200005000-00004. PMID 11256663
- [Background] Centers for Disease Control and Prevention (CDC). Awareness of family health history as a risk factor for disease--United States, 2004. MMWR Morb Mortal Wkly Rep. 2004 Nov 12;53(44):1044-7. PMID 15538320
- [Background] Qureshi N, Wilson B, Santaguida P, Carroll J, Allanson J, Culebro CR, Brouwers M, Raina P. Collection and use of cancer family history in primary care. Evid Rep Technol Assess (Full Rep). 2007 Oct;(159):1-84. PMID 18457477
- [Background] Wagner EH, Austin BT, Von Korff M. Organizing care for patients with chronic illness. Milbank Q. 1996;74(4):511-44. PMID 8941260
- [Background] Glasgow RE, McKay HG, Piette JD, Reynolds KD. The RE-AIM framework for evaluating interventions: what can it tell us about approaches to chronic illness management? Patient Educ Couns. 2001 Aug;44(2):119-27. doi: 10.1016/s0738-3991(00)00186-5. PMID 11479052
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Acheson LS, Zyzanski SJ, Stange KC, Deptowicz A, Wiesner GL. Validation of a self-administered, computerized tool for collecting and displaying the family history of cancer. J Clin Oncol. 2006 Dec 1;24(34):5395-402. doi: 10.1200/JCO.2006.07.2462. Epub 2006 Nov 6. PMID 17088568
- [Background] Scheuner MT, Wang SJ, Raffel LJ, Larabell SK, Rotter JI. Family history: a comprehensive genetic risk assessment method for the chronic conditions of adulthood. Am J Med Genet. 1997 Aug 22;71(3):315-24. doi: 10.1002/(sici)1096-8628(19970822)71:33.0.co;2-n. PMID 9268102
- [Background] Karliner LS, Napoles-Springer A, Kerlikowske K, Haas JS, Gregorich SE, Kaplan CP. Missed opportunities: family history and behavioral risk factors in breast cancer risk assessment among a multiethnic group of women. J Gen Intern Med. 2007 Mar;22(3):308-14. doi: 10.1007/s11606-006-0087-y. PMID 17356960
- [Background] Kaplan CP, Haas JS, Perez-Stable EJ, Gregorich SE, Somkin C, Des Jarlais G, Kerlikowske K. Breast cancer risk reduction options: awareness, discussion, and use among women from four ethnic groups. Cancer Epidemiol Biomarkers Prev. 2006 Jan;15(1):162-6. doi: 10.1158/1055-9965.EPI-04-0758. PMID 16434605
- [Background] Murff HJ, Byrne D, Haas JS, Puopolo AL, Brennan TA. Race and family history assessment for breast cancer. J Gen Intern Med. 2005 Jan;20(1):75-80. doi: 10.1111/j.1525-1497.2004.40112.x. PMID 15693932
- [Background] Weingart SN, Hamrick HE, Tutkus S, Carbo A, Sands DZ, Tess A, Davis RB, Bates DW, Phillips RS. Medication safety messages for patients via the web portal: the MedCheck intervention. Int J Med Inform. 2008 Mar;77(3):161-8. doi: 10.1016/j.ijmedinf.2007.04.007. Epub 2007 Jun 19. PMID 17581772
- [Background] Adler-Milstein J, Bates DW, Jha AK. U.S. Regional health information organizations: progress and challenges. Health Aff (Millwood). 2009 Mar-Apr;28(2):483-92. doi: 10.1377/hlthaff.28.2.483. PMID 19276008
- [Background] Wright A, Poon EG, Wald J, Schnipper JL, Grant R, Gandhi TK, Volk LA, Bloom A, Williams DH, Gardner K, Epstein M, Nelson L, Businger A, Li Q, Bates DW, Middleton B. Effectiveness of health maintenance reminders provided directly to patients. AMIA Annu Symp Proc. 2008 Nov 6:1183. PMID 18999087
- [Background] Linder JA, Ma J, Bates DW, Middleton B, Stafford RS. Electronic health record use and the quality of ambulatory care in the United States. Arch Intern Med. 2007 Jul 9;167(13):1400-5. doi: 10.1001/archinte.167.13.1400. PMID 17620534
- [Background] Ozanne EM, Loberg A, Hughes S, Lawrence C, Drohan B, Semine A, Jellinek M, Cronin C, Milham F, Dowd D, Block C, Lockhart D, Sharko J, Grinstein G, Hughes KS. Identification and management of women at high risk for hereditary breast/ovarian cancer syndrome. Breast J. 2009 Mar-Apr;15(2):155-62. doi: 10.1111/j.1524-4741.2009.00690.x. PMID 19292801
- [Background] Dominguez FJ, Lawrence C, Halpern EF, Drohan B, Grinstein G, Black DM, Smith BL, Gadd MA, Specht M, Kopans DB, Moore RH, Hughes SS, Roche CA, Hughes KS. Accuracy of self-reported personal history of cancer in an outpatient breast center. J Genet Couns. 2007 Jun;16(3):341-5. doi: 10.1007/s10897-006-9067-y. Epub 2007 May 17. PMID 17508275
- [Background] Guttmacher AE, Collins FS, Carmona RH. The family history--more important than ever. N Engl J Med. 2004 Nov 25;351(22):2333-6. doi: 10.1056/NEJMsb042979. No abstract available. PMID 15564550